CLINICAL TRIAL: NCT04639193
Title: Rescuing OSA Patients Unable to Tolerate CPAP Using Endotype-Targeted Combination Drug Therapy: a Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Combination Drug-Therapy for Patients With Untreated Obstructive Sleep Apnea
Acronym: RESCUE-Combo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Principal Investigator, Christopher Schmickl, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191990
Record Dates: First submitted 2020-11-12; First posted 2020-11-20 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: OSA; Obstructive Sleep Apnea
Keywords: sleep; drug
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide; Eszopiclone; Venlafaxine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo, then Dual-Therapy, then Single/Triple-Therapy (Experimental): Subjects will start with a 3-day PLACEBO regimen:
  * Day 1: Placebo (matching Acetazolamide 250mg) at bedtime at home.
  * Day 2: Placebo (matching Acetazolamide 500mg) at bedtime at home.
  * Day 3: Placebo (matching Acetazolamide 500mg + Eszopiclone 2mg) at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects will then cross-over to a 3-day EXPERIMENTAL DUAL-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects will then undergo an OPEN-LABEL SINGLE/TRIPLE-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg alone or Acetazolamide 500mg + Eszopiclone 2mg + Venlafaxine 50mg at bedtime in the sleep laboratory, if sleep apnea resolved or did not resolve with the dual regimen, respectively.
  Interventions: Drug: Acetazolamide; Drug: Eszopiclone; Drug: Placebo; Drug: Venlafaxine
- Dual-Therapy, then Placebo, then Single/Triple-Therapy (Experimental): Subjects will start with a 3-day EXPERIMENTAL DUAL-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects will then cross-over to a 3-day PLACEBO regimen:
  * Day 1: Placebo (matching Acetazolamide 250mg) at bedtime at home.
  * Day 2: Placebo (matching Acetazolamide 500mg) at bedtime at home.
  * Day 3: Placebo (matching Acetazolamide 500mg + Eszopiclone 2mg) at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects will then undergo an OPEN-LABEL SINGLE/TRIPLE-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg alone or Acetazolamide 500mg + Eszopiclone 2mg + Venlafaxine 50mg at bedtime in the sleep laboratory, if sleep apnea resolved or did not resolve with the dual regimen, respectively.
  Interventions: Drug: Acetazolamide; Drug: Eszopiclone; Drug: Placebo; Drug: Venlafaxine

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide tablet (encapsulated)
  Other Names: Diamox
Drug: Eszopiclone — Eszopiclone tablet (encapsulated)
  Other Names: Lunesta
Drug: Placebo — Sugar capsule manufactured to match encapsulated Acetazolamide/Eszopiclone
Drug: Venlafaxine — Venlafaxine capsule
  Other Names: Effexor

SUMMARY:
Obstructive sleep apnea (OSA) is common and associated with many adverse health consequences, but many patients are unable to tolerate standard therapies such as continuous positive airway pressure (CPAP) and thus remain untreated. Single-drug therapies have shown promising results in treating sleep apnea, but on average patients have only experienced partial relief. Multi-drug therapy may offer a more effective treatment approach. The goal of this study is to test the effect of combination therapy with three FDA-approved drugs (Diamox [acetazolamide], Lunesta [eszopiclone] +/- Effexor [venlafaxine]) on OSA severity and physiology.

DETAILED DESCRIPTION:
Study participants will undergo three 3-day drug regimens. On days 1 and 2 of each drug regimen, subjects will take the study drugs at home; on day 3 of each drug regimen subjects will take the study drugs as part of an overnight inlab sleep study (including assessments of sleepiness/alertness, sleep quality and blood pressure). Initially subjects will take dual-therapy (acetazolamide+eszopiclone) vs placebo in random order; if sleep apnea resolved with dual-therapy, then subjects will undergo an open-label single-drug regimen (acetazolamide), else an open-label triple-drug regimen (acetazolamide + eszopiclone + venlafaxine).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-40 kg/m2
* Untreated Moderate or Severe OSA (AHI during supine NREM sleep >15/h) with a fraction of hypopneas >25% of all events

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Prisoners
* Adherent with effective therapy for OSA
* Other known untreated sleep fragmenting disorder, such as periodic limb movement disorder, or narcolepsy
* Inability to sleep supine for overnight sleep studies
* Circadian rhythm disorder
* Unrevascularized coronary artery disease, angina, prior heart attack or stroke, congestive heart failure
* Uncontrolled hypertension (systolic blood pressure >160mmHg, diastolic blood pressure >95mmHg)
* Presence of tracheostomy
* Hospitalization within the past 90 days
* Prior peptic ulcer disease, esophageal varices, or gastrointestinal bleeding (< 5 years)
* Prior gastric bypass surgery
* Chronic liver disease or end-stage kidney disease
* Active illicit substance use or >2 oz daily alcohol use (i.e. >2 12 oz bottles of beers, >2 5 oz glasses of wine, >2 1.5 oz glasses of hard liquor such as spirits, gin, whiskey, etc.)
* Psychiatric disease, other than well controlled depression/anxiety
* Cognitive impairment, inability to provide consent, or inability to complete research procedures (e.g. questionnaires that are only available/validated in English)
* Chronically using study drugs or drugs with similar pharmacodynamic effects (acetazolamide - carbonic anhydrase inhibitors, eszopiclone - benzodiazepine receptor agonists, venlafaxine - serotonin/norepinephrine reuptake inhibitors and other antidepressants)
* Regular use of medications known to affect control of breathing (opioids, benzodiazepines, theophylline)
* Contraindications to taking study drugs, including allergies to any of the drugs or sulfa allergy; concomitant use of antidepressants, opioids, sedatives/hypnotics, thiazide diuretics or angiotensin-receptor blockers; or severe nocturnal hypoxia (SpO2 nadir <70% on diagnostic sleep study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schmickl, MD, PhD, Principal Investigator — Associate Physician and Postdoctoral Fellow
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute Building, La Jolla, California
  - UCSD Health - Pulmonary and Sleep Clinic, La Jolla, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmickl CN, Orr JE, Alex RM, Gruenberg E, Parra G, White S, Spenceley A, DeSarkar T, Kong M, DeYoung PN, Sands SA, Owens RL, Malhotra A. Combination Drug Therapy with Acetazolamide, Eszopiclone +/- Venlafaxine for Obstructive Sleep Apnea (RESCUE-Combo): A Randomized, Double-Blind, Placebo-controlled Clinical Trial. Ann Am Thorac Soc. 2025 Feb;22(2):263-273. doi: 10.1513/AnnalsATS.202407-736OC. PMID 39514000

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 88 subjects who were assessed for eligibility, 20 were randomized. The other 68 were excluded due to not meeting eligibility criteria or not being interested.
Groups:
- Placebo, Then Dual-Therapy, Then Triple-Therapy: Subjects started with a 3-day PLACEBO regimen:
  * Day 1: Placebo (matching Acetazolamide 250mg) at bedtime at home.
  * Day 2: Placebo (matching Acetazolamide 500mg) at bedtime at home.
  * Day 3: Placebo (matching Acetazolamide 500mg + Eszopiclone 2mg) at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects then crossed over to a 3-day EXPERIMENTAL DUAL-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects then underwent an OPEN-LABEL TRIPLE-regimen:
  Day 1: Acetazolamide 250mg at bedtime at home. Day 2: Acetazolamide 500mg at bedtime at home. Day 3: Acetazolamide 500mg + Eszopiclone 2mg + Venlafaxine 50mg at bedtime in the sleep laboratory
  Acetazolamide: Acetazolamide tablet (encapsulated) Eszopiclone: Eszopiclone tablet (encapsulated) Placebo: Sugar capsule manufactured to match encapsulated Acetazolamide/Eszopiclone Venlafaxine: Venlafaxine capsule
- Dual-Therapy, Then Placebo, Then Triple-Therapy: Subjects started with a 3-day EXPERIMENTAL DUAL-regimen:
  * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects then crossed over to a 3-day PLACEBO regimen:
  * Day 1: Placebo (matching Acetazolamide 250mg) at bedtime at home.
  * Day 2: Placebo (matching Acetazolamide 500mg) at bedtime at home.
  * Day 3: Placebo (matching Acetazolamide 500mg + Eszopiclone 2mg) at bedtime in the sleep laboratory.
  After a wash-out period of 4+ days, subjects then underwent an OPEN-LABEL TRIPLE-regimen:
  Day 1: Acetazolamide 250mg at bedtime at home. Day 2: Acetazolamide 500mg at bedtime at home. Day 3: Acetazolamide 500mg + Eszopiclone 2mg + Venlafaxine 50mg at bedtime in the sleep laboratory
  Acetazolamide: Acetazolamide tablet (encapsulated) Eszopiclone: Eszopiclone tablet (encapsulated) Placebo: Sugar capsule manufactured to match encapsulated Acetazolamide/Eszopiclone Venlafaxine: Venlafaxine capsule
Period: First Intervention
Arm/Group | Placebo, Then Dual-Therapy, Then Triple-Therapy | Dual-Therapy, Then Placebo, Then Triple-Therapy
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo, Then Dual-Therapy, Then Triple-Therapy | Dual-Therapy, Then Placebo, Then Triple-Therapy
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | Placebo, Then Dual-Therapy, Then Triple-Therapy | Dual-Therapy, Then Placebo, Then Triple-Therapy
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Who Were Enrolled Into the Trial: All 20 participants who were randomized, completed the dual-therapy and placebo phases (blinded/random order) 18 of these 20 participants went on to also complete the the open label triple therapy phase
Arm/Group | All Participants Who Were Enrolled Into the Trial
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [36 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 29.1 [27.6 to 34.2]
Apnea Hypopnea Index (AHI) [Median (Inter-Quartile Range); unit: events/hour of sleep] — The AHI is a measure of sleep apnea severity and is defined as the number of apneas (no breathing for 10+ seconds) and hypopneas (reduced breathing for 10+ seconds associated with a >=3% desaturation or cortical arousal) per hour of sleep. To avoid confounding by sleep stages and positions across study nights the primary focus was on the AHI during supine non rapid eye movement (NREM) sleep. The "AHI4" defines hypopneas as reduced breathing for 10+ seconds associated with a >=4% desaturation.
  events/hour of sleep
    AHI (supine, NREM) | 32.8 [20 to 48.8]
    AHI (overall) | 39.2 [21.5 to 50.7]
    AHI4 (overall) | 21.8 [10.8 to 29.9]
Pathophysiological Traits: Vpassive, Vactive, Arousal Threshold [Median (Inter-Quartile Range); unit: % Veupnea] — Pathophysiological traits were quantified as %Veupnea from polysomnography data using a validated algorithm.
  % Veupnea
    Vpasssive, transformed | 69.9 [61.1 to 73]
    Vactive | 92.1 [79.2 to 97.9]
    Arousal Threshold, transformed | 142 [127.7 to 156.1]
Pathophysiological Trait: Loop Gain [Median (Inter-Quartile Range); unit: dimensionless] — Loop Gain 1 was quantified from polysomnography data using a validated algorithm. This metric measures the increase in respiratory drive relative to a preceding drop in ventilation and thus is dimensionless (typical range is approximately 0.2 to 1.5, with values >0.7 being considered high loop gain, indicating ventilatory instability).
  dimensionless | 0.56 [0.50 to 0.65]

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: The AHI is a measure of sleep apnea severity and based on the American Academy of Sleep Medicine (AASM)-recommended criteria is defined as the number of apneas (no breathing for 10+ seconds) and hypopneas (reduced breathing for 10+ seconds associated with a >=3% desaturation or cortical arousal) per hour of sleep. To avoid confounding by sleep stages and positions across study nights the primary focus was on the AHI during supine non rapid eye movement (NREM) sleep. For comparability with other studies, we also explored the AASM-acceptable "AHI4", which defines hypopneas as reduced breathing for 10+ seconds associated with a >=4% desaturation.
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: events/hour of sleep
Groups:
- Dual-Therapy: * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg at bedtime in the sleep laboratory.
- Placebo: * Day 1: Placebo (matching Acetazolamide 250mg) at bedtime at home.
  * Day 2: Placebo (matching Acetazolamide 500mg) at bedtime at home.
  * Day 3: Placebo (matching Acetazolamide 500mg + Eszopiclone 2mg) at bedtime in the sleep laboratory.
- Triple-Therapy: * Day 1: Acetazolamide 250mg at bedtime at home.
  * Day 2: Acetazolamide 500mg at bedtime at home.
  * Day 3: Acetazolamide 500mg + Eszopiclone 2mg + Venlafaxine 50mg at bedtime in the sleep laboratory.
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
events/hour of sleep
  AHI (supine, NREM) | 17.1 [9.4 to 37.7] | 32.7 [23.8 to 51.8] | 26 [9.2 to 40]
  AHI (overall) | 23.6 [15.2 to 38.3] | 37.4 [30.4 to 50] | 25.8 [9.9 to 43.3]
  AHI4 (overall) | 14.1 [7.9 to 27.3] | 20.3 [13.3 to 37.9] | 9 [4.5 to 14.7]

2. Secondary Outcome: SpO2 Nadir
Description: The lowest measured blood oxygen saturation during the overnight sleep study measured in percent.
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: Percent Oxygen Saturation
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
Percent Oxygen Saturation | 83.5 [79.8 to 87.2] | 84 [82 to 85.2] | 86 [82.5 to 87.5]

3. Secondary Outcome: Pathophysiological Traits: Vpassive, Vactive, Arousal Threshold
Description: Pathophysiological traits were quantified as %Veupnea from polysomnography data using a validated algorithm.
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: % Veupnea
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
% Veupnea
  Vpasssive, transformed | 69.5 [58.7 to 78.2] | 67.4 [59.4 to 73.2] | 70.4 [61.7 to 75.3]
  Vactive | 96.2 [79 to 99.1] | 92.1 [83.9 to 97.7] | 94.4 [83.9 to 99.6]
  Arousal Threshold, transformed | 140.1 [126.7 to 161.5] | 149.8 [137.9 to 162.2] | 137.2 [125 to 155.7]

4. Secondary Outcome: Pathophysiological Trait: Loop Gain
Description: Loop Gain 1 was quantified from polysomnography data using a validated algorithm. This metric measures the increase in respiratory drive relative to a preceding drop in ventilation and thus is dimensionless (typical range is approximately 0.2 to 1.5, with values >0.7 being considered high loop gain, indicating ventilatory instability)
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: dimensionless
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
dimensionless | 0.54 [0.49 to 0.59] | 0.57 [0.51 to 0.69] | 0.49 [0.44 to 0.6]

5. Secondary Outcome: Percent Responders
Description: Full responders were defined as a drop in AHI>50% to <10/h.
Time Frame: 3 nights
Measure: Count of Participants; unit: Participants
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
Participants
  Based on AHI in supine NREM sleep | 5 | 0 | 4
  Based on AHI overall | 1 | 1 | 4

6. Secondary Outcome: Blood Pressure
Description: Systolic/Diastolic Blood Pressure (measured at rest in the morning following the overnight sleep study).
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
mmHg
  Systolic Blood Pressure | 112.5 [107.8 to 119.8] | 116.5 [109.8 to 124.5] | 116 [110.2 to 120.8]
  Diastolic Blood Pressure | 72 [67.8 to 78.2] | 74 [68.5 to 82] | 70.5 [63.2 to 79.5]

7. Secondary Outcome: Subjective Sleepiness: Stanford Sleepiness Scale (SSS)
Description: Subjective sleepiness was assessed using the Stanford Sleepiness Scale (SSS) in the morning following the overnight sleep study. The score ranges from 1 to 7, with greater values indicating more sleepiness.
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
units on a scale | 2 [1 to 2.2] | 2 [1 to 3] | 2 [1 to 3.8]

8. Secondary Outcome: Sleep Quality: PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance
Description: Sleep quality was assessed based on a modified 8-question PROMIS Sleep Disturbance (SDA 8b) questionnaire in the morning following the overnight sleep study. The raw score ranges from 8 to 40 and is translated into a T-score, a standardized score with a mean of 50 and a standard deviation of 10. Greater T-scores indicate greater sleep disturbance.
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: t-score
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
t-score | 53 [49 to 56.3] | 53.9 [49.9 to 57.8] | 53 [48.8 to 55.6]

9. Secondary Outcome: Psychomotor Vigilance: Response Speed
Description: Vigilance was assessed using the 10-minute psychomotor vigilance test (PVT) in the morning following the overnight sleep study. Primary focus was on "response speed" 1/reaction time (1/RT) and lapses (reaction time >500ms).
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: 1/seconds
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
1/seconds | 3 [2.8 to 3.3] | 3.1 [2.8 to 3.4] | 2.9 [2.8 to 3.3]

10. Secondary Outcome: Psychomotor Vigilance: Lapses
Description: as for outcome 9
Time Frame: 3 nights
Measure: Median (Inter-Quartile Range); unit: Number of lapses
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
Number analyzed (Participants) | 20 | 20 | 18
Number of lapses | 3 [0 to 8.2] | 3 [1 to 6.2] | 5 [2.2 to 9.8]

ADVERSE EVENTS:
Time Frame: During the trial subjects were asked at each visit whether any adverse events had occurred during that 3-day study phase.
Arm/Group | Dual-Therapy | Placebo | Triple-Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 11/20 | 10/20 | 16/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dual-Therapy (N=20) | Placebo (N=20) | Triple-Therapy (N=18)
Bad Dreams (General disorders) | 1 | 0 | 0
Cloudy Urine (Renal and urinary disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Abnormal Taste when Drinking Carbonated Beverages (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 1 | 0
Gastrointestinal Upset (Gastrointestinal disorders) | 0 | 0 | 6
Hand Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (General disorders) | 0 | 0 | 2
Heartburn (Gastrointestinal disorders) | 0 | 0 | 1
Hot Flashes (General disorders) | 0 | 1 | 0
Itchiness (General disorders) | 0 | 1 | 0
Metallic Taste (General disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 3 | 0 | 2
Polyuria (Renal and urinary disorders) | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Shoulder Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sleepiness (General disorders) | 5 | 4 | 8
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04639193/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04639193/ICF_001.pdf